CLINICAL TRIAL: NCT01307657
Title: Impact of a High-fat Meal on Assessment of Clopidogrel-induced Platelet Inhibition in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0568-10-FB
Record Dates: First submitted 2011-02-22; First posted 2011-03-03 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Healthy
Keywords: clopidogrel; platelet; platelet function test; healthy; Platelet function tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clopidogrel impact on platelet function (Other): Participants will have a baseline blood sample drawn after a 12 hour fast at 8 am, then be administered a 600 mg dose of clopidogrel. At noon, another blood sample will be drawn to evaluate the extent of maximum platelet inhibition in the fasting state. Participants will then be provided a standardized high-fat meal, then an additional blood sample at 2 pm to evaluate the impact of the high-fat on platelet function assessment.
  Interventions: Other: high fat meal

INTERVENTIONS:
Other: high fat meal — Clopidogrel 600 mg loading dose at 8 am and high-fat meal at 12 pm

SUMMARY:
The purpose of this study is to determine whether a high-fat meal affects the ability of platelet function tests to measure platelet inhibition by clopidogrel.

DETAILED DESCRIPTION:
The purpose of this study is to determine the influence of a high-fat meal on assessment of clopidogrel-induced platelet inhibition in healthy people using platelet function assays. Twelve healthy adult subjects will be recruited to take part in this research study. After consent is obtained, subjects will be asked to present to the clinical research center after a 12 hour fast. A baseline blood sample will be drawn at 8 am, and subjects will then be administered a 600 mg dose of clopidogrel. At 12 noon, another blood sample will be drawn to evaluate the extent of maximum platelet inhibition in the fasting state. Subjects will then be provided a standardized high-fat meal with an additional blood sample at 2 pm to evaluate the impact of the high-fat on platelet function assessment.

ELIGIBILITY:
Inclusion Criteria:

* 19 years of age or older
* healthy subjects
* deny taking medications that affect platelet function for at least 7 days prior to test

Exclusion Criteria:

* history of cardiovascular disease
* any risk factors for cardiovascular disease
* surgery in last 3 months
* history of anemia/thrombocytopenia
* pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-02-15 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2012-03-01 (Actual)

PRIMARY OUTCOMES:
Platelet inhibition | 3 time points over 6 hours
  platelet inhibition before versus after a high-fat meal (measured by light transmission aggregometry, whole blood aggregometry, flow cytometry, and VerifyNow assay)

CONTACTS AND LOCATIONS:
Overall Officials: Julie Oestreich, PharmD, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Dobesh PP, Urban JF, Shurmur SW, Oestreich JH. Impact of a high-fat meal on assessment of clopidogrel-induced platelet inhibition in healthy subjects. Thromb J. 2015 Jan 23;13(1):3. doi: 10.1186/s12959-014-0033-x. eCollection 2015. PMID 25642145